CLINICAL TRIAL: NCT01583712
Title: Diagnosis of Acute Gastrointestinal Graft-versus-Host Disease by Early Endomicroscopic Features of the Small Intestine
Brief Title: Endomicroscopy and Graft-versus-host Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Prinicpal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 787/2010
Record Dates: First submitted 2012-01-08; First posted 2012-04-24 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Haematopoietic Stem Cell Transplantation
Keywords: Confocal laser endomicroscopy; Small bowel imaging; Graft-versus-host disease; HSCT
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endomicroscopy (Experimental): All patients included in the study will undergo endomicroscopy of the upper GI-tract including the reachable parts of the small bowel.
  Interventions: Procedure: Confocal laser endomicroscopy; Device: Confocal Laser Endomicroscope

INTERVENTIONS:
Procedure: Confocal laser endomicroscopy — Endomicroscopy of the upper gastrointestinal tract including endomicroscopic pictures taken every ten centimetres in the small bowel, gastric antrum, gastric corpus and esophagus.
Device: Confocal Laser Endomicroscope — Pentax EC-3870 CIFK with the ISC-1000 confocal endomicroscopy processor - Pentax, Tokyo, Japan and Optiscan Pty Ltd, Notting Hill, Victoria, Australia

SUMMARY:
Early diagnosis of acute Gastrointestinal Graft-versus-Host disease (aGI-GvHD) has a strong impact on morbidity and mortality of patients who underwent haematopoietic stem cell transplantation (HSCT). Recent results at the investigators department showed that mucosal biopsies from the small intestine have a high diagnostic yield for aGI-GvHD specific changes. By performing an enteroscopic examination, aGI-GvHD suspected patients can be prevented from colonoscopy and prior bowel preparation which is clinically important, considering the rather bad general condition of this patient group. To further reduce invasive procedures the investigators want to evaluate the in vivo histological features of aGI-GvHD in the small bowel. Therefore aGI-GvHD suspected patients will undergo confocal laser endomicroscopy of the upper GI-tract, including duodenum and jejunum, in the context of a prospective clinical pilot trial. The histological evaluation of biopsy samples taken from these sites will be used as comparable gold standard. Endomicroscopic aspects of patients with celiac disease, infectious enteritis, inflammatory bowel disease and healthy subjects should serve as controls. If it is possible to diagnose aGI-GvHD from endomicroscopic features of the small bowel alone, this could be another important step to improve the diagnostic management of post HSCT patients, especially when taking of biopsy samples is difficult because of a bad coagulation status. Additionally, an accurate diagnosis in vivo could lead to immediate treatment to prevent progression and site spreading of the disease.

DETAILED DESCRIPTION:
Graft-versus-host disease (GvHD) represents a major cause for morbidity and mortality in patients who underwent haematopoietic stem cell transplantation (HSCT) [1]. In the gastrointestinal tract as one of the main target organs of GvHD diagnosis may be difficult because of many similar presenting differential diagnoses, most notable, infections by cytomegalovirus [2]. Experts disagree about the best diagnostic approach for patients suspected of acute gastrointestinal GvHD (aGI-GvHD). There have been many studies supporting the endoscopic evaluation of either the lower [3, 4, 5], the upper [6, 7] or both parts of the GI-tract [8, 9]. In either case, the histological evaluation of biopsy samples serves as standard tool to establish the final diagnosis [10].

Considering the rather bad general condition of patients after HSCT as a limiting factor for endoscopic and histological evaluation, some new approaches have been introduced into the diagnostic manual of aGI-GvHD in order to reduce the amount of invasive examinations. Conventional imaging techniques like magnetic resonance imaging [11], computer tomography [12] and high-resolution ultrasonography with Doppler Imaging [13] reported bowel wall thickening in GvHD patients. But as such findings are only unspecific signs of gastrointestinal pathology, conventional imaging techniques cannot replace endoscopy with biopsies [14]. The same holds for video capsule endoscopy which was indeed found to have a high negative predictive value for the detection of aGI-GvHD, but shares the important shortcoming of missing biopsy samples for histological evaluation [15, 16, 17].

At least this method shifted the focus of interest onto the small bowel. Biopsies deriving from this former neglected GI part had shown a high sensitivity for GvHD-related changes in previous studies [18]. As similar results were seen at the study site, the investigators prospectively compared enteroscopy with biopsies to the present gold standard in the diagnostic aGI-GvHD management, colonoscopy with biopsies. In the context of this investigation the large intestine showed much stronger affection by aGI-GvHD than all other locations, although there was no pair of examinations, in which colonoscopy revealed aGI-GvHD without the presence of such findings at enteroscopy. Quite the opposite, enteroscopy even revealed GvHD related pathologies in one case where the respective colonoscopy remained inconspicuous. Consequently, they postulated that enteroscopic findings may replace the need for colonoscopy [19], wherefore post-HSCT patients could remain without stressful bowel preparation, often limited by their rather bad general condition.

One of the latest developments in the endoscopic management of the gastrointestinal tract is the so called confocal laser endomicroscope (CLE). Confocal microscopy was developed by Marvin Minsky in the late 1950s. Its principle is the microscopic scanning of focal points below the surface of an object. In comparison to conventional light microscopy it uses a special filter system to avoid image overlapping by surrounding tissue. In detail, a light source (normally a laser) is focused by a microscope objective lens to a diffraction limited spot on or inside the object. Light that is scattered, or fluorescence excited (achieved through fluorescein staining, for example) and emitted, at the focus in the sample will partially return back through the optics along the path from which it arrived. A beam-splitter placed into the path reflects the return light towards a detector. The optics will focus the light from the focal point in the specimen to its conjugate focus near the detector (hence the technology is termed "con-focal"). Here a spatial filter ("pinhole") is used to extinguish all light deriving from areas outside the focal point. Light reflections from the focal point itself will be forwarded to the detector which is connected to a computer system that digitalises the optical signal and creates the in vivo histological image [20].

Focusing on its clinical impact, confocal microscopy is the first technique to allow in vivo evaluation of tissue structures beneath their surface. Because of many breakthroughs in miniaturisation (mostly in the 1990s) this technology could be applied for intraluminal use in gastroenterology, integrated into a otherwise standard endoscope. It allows the in vivo histological visualisation of the upper 250 micrometers of all walls within the gastrointestinal tract, additionally to the normal function of white light endoscopy (provided by two separate screens on top of the workstation) [20].

The first clinical use of CLE in a prospective pilot trial including 35 patients after HSCT was reported by Bojarski et al. in 2009. CLE of the colonic mucosa could predict the positive diagnosis of aGI-GvHD in 14 of 19 patients, later confirmed by histological evaluation. The in vivo findings of aGI-GvHD, varying from single crypt apoptosis to complete crypt loss, were clearly distinguishable from pathologies of other origin like infectious colitis or ulcerative colitis, both used as comparative control [21].

Study Aims

In this clinical investigation the investigators intend to continue the diagnostic approach for acute Gastrointestinal Graft-versus-Host Disease (aGI-GvHD). Based on the recent results at the study institution (explained above, [19]) that showed a remarkable diagnostic yield for aGI-GvHD associated pathologies in the small intestine the investigators intend to evaluate confocal laser endomicroscopy (CLE) of the small intestine as primary diagnostic procedure in patients with suspected aGI-GvHD after haematopoietic stem cell transplantation (HSCT).

* The investigators aim to examine whether early diagnosis of aGI-GvHD in the duodenum and jejunum can be achieved by evaluating endomicroscopic features.
* In comparison with conventional biopsies from the mentioned GI-parts as gold standard the investigators want to test whether the markers described by Bojarski et al. for the colon also hold true for the small intestine.
* Including endomicroscopic results of patients with celiac disease, enteral infections, inflammatory bowel disease and healthy subjects as controls the investigators aim to establish aGI-GvHD specific markers that can be used for a "biopsy-free" in vivo diagnosis of aGI-GvHD.

Study Design

Prospective clinical pilot trial without randomisation or blinding

Study Population

Patients after haematopoietic stem cell transplantation (HSCT) who are referred to the study site for clarification of one of the following symptoms:

* anorexia
* nausea
* vomiting
* abdominal pain
* diarrhea
* intestinal bleeding

To exclude possible side effects of the conditioning therapy, GI symptoms must have occurred or persisted 20 days after the respective transplantation date [22].

Exclusion criteria:

* infection with CMV or HSV
* bacterial infection of the GI tract
* medication related symptoms
* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* refusal to participate in the study
* patient's age below 18 years.

Methods

This investigation will be performed at the Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology. Patient recruitment will be achieved in close cooperation with the Department of Internal Medicine I, Division of Oncology, Bone Marrow Transplantation Unit.

As this study has been planned as a pilot trial, it mainly focuses on the qualitative endomicroscopic features of the small intestine in GvHD-patients to yield reference pathologies for accurate diagnosis in the future. Nevertheless, a quantitative analysis will be performed by comparing CLE-derived diagnoses with histological results to calculate sensitivity and specificity of CLE-based aGI-GvHD diagnosis in the small intestine. Considering the current diagnostic yield of 62% for the detection of aGI-GvHD in symptomatic post-HSCT-patients by conventional histology [19], the investigators estimated to include 40 patients with suspected aGI-GvHD in order to discover a meaningful sample of patients affected by aGI-GvHD for qualitative and quantitative analysis. In comparison, Bojarski et al included 35 patients of whom 19 finally turned out to suffer from aGI-GvHD by conventional histology. They could then calculate a sensitivity of 74% and specificity of 100% for the prediction of the histological diagnosis by CLE [21]. On the basis of the current frequency of post-HSCT-patients at the study site the investigators estimate to include the aimed amount of 40 patients within a time period of 2 years.

All patients who fulfill the listed inclusion criteria, will receive the patient information form of this study together with the usual informed consent form of the respective endoscopic examination they are about to undergo. Patient information will be done at least 24 hours before the intervention, as practiced at our unit. If the patient agrees to participate in the study he/she will be prepared for endoscopy by administration of intravenous propofol and/or midazolam as routinely used for conscious sedation during endoscopic procedures at our department. Additionally, 5-10 ml of a 10% solution of fluorescein sodium will be administered intravenously to enhance tissue fluorescence during endomicroscopy. As so far no specific CLE-enteroscope is available, we will use the CLE-colonoscope (Pentax EC-3870 CIFK with the ISC-1000 confocal endomicroscopy processor - Pentax, Tokyo, Japan and Optiscan Pty Ltd, Notting Hill, Victoria, Australia) to reach the small intestine, comparable to an enteroscopic procedure (oral access).

All drugs will be administered by medical specialists, assistant doctors or registered nurses, as routinely practiced at our institution.

CLE picture capturing will start at the deepest point reachable in the jejunum. During withdrawal of the scope CLE pictures will be taken every 10 centimetres in the small bowel, then from the antrum and body of the stomach and from the esophagus. Furthermore, CLE will be applied for distinct looking areas, suspicious of pathologic origin. Wherever CLE pictures are obtained, a conventional biopsy will be taken from the same localisation.

CLE pictures will be captured and stored routinely using our standard data management system. They will be evaluated immediately after the endoscopic procedure together with a board certified GI-pathologist, who will establish an initial diagnosis.

Conventional biopsies will be stained with Haematoxylin & Eosin, as well as PAS stain. In-situ hybridization for CMV and HSV will be performed to exclude viral infection. Classification of GvHD will be done according to McDonald and Sale in 4 grades, appropriately modified for the small intestine [23]:

* Grade I: individual cell necrosis
* Grade II: crypt abscess
* Grade III: drop out of one ore more whole crypts in a biopsy
* Grade IV: total denudation of epithelium

Endomicroscopic controls (patients with celiac disease, enteral infections, inflammatory bowel disease and healthy subjects) will be collected from present data of endomicroscopic procedures already performed within routine examinations.

At the end of the study all CLE pictures and histological cuts will be evaluated separately by two blinded board certified pathologists. In case of discordant diagnoses they will analyse the respective cases together to reach an agreement on the final diagnosis. All cases where the initial and the final diagnosis are deviating from each other will be re-evaluated together by all specialists involved.

Risk/Benefit assessment

GvHD represents a major cause of morbidity and mortality after allogeneic HSCT. Approximately 10-40% of patients who undergo HSCT develop significant GvHD, and about half of these patients die from this disease or from therapy resulting complications [1].

Endoscopic procedures in patients with suspected aGI-GvHD are well established. Until now the histological evaluation of GI deriving biopsies is the gold standard tool to set an accurate aGI-GvHD diagnosis. Endoscopy of the upper GI-tract is more comfortable than the endoscopic assessment of the lower GI-tract as there is no need for bowel preparation. Therefore it is the primary technique to assess post HSCT patients at our department. Supported by recent results at the study institution [19] these upper GI endoscopies are routinely performed as enteroscopies instead of gastroscopies in order to include the small intestine in the diagnostic evaluation. The safety of enteroscopy has not been studied systematically but reported experience is substantial and complications have been rare [24].

Confocal laser endomicroscopy is a safe new technique that has already been studied in clinical trials [25, 26]. Its safety is being guaranteed by the use of low intensity laser light that can at worst cause local bleaching of fluorescein containing cells, which is harmless, reversible and even used as diagnostic sign in experimental conditions [20].

Ethical implications

This study protocol was approved by the ethics commission of the Medical University of Vienna.

All procedures in the context of this study will be performed in accordance to the Declaration of Helsinki as well as to the guidelines for Good Scientific Practice (GSP) of the Medical University of Vienna.

Expected impact and Outlook

If the investigators find aGI-GvHD specific markers that can be used for a "biopsy-free" in vivo diagnosis of aGI-GvHD this could lead to another reduction of invasive procedures for patients after HSCT. This would have a big clinical impact, as biopsy assessment is often limited by the bad coagulation status of this patient group.

In case they cannot clearly determine specific markers of aGI-GvHD, CLE should at least reduce the amount of conventional biopsies needed for diagnosis by taking them under CLE guidance.

Despite from the expected reduction of invasive procedures, aGI-GvHD diagnosis in vivo could lead to immediate initiation of immunosuppressive treatment in order to reduce progression and site spreading of the disease.

In case the study aims will be supported by the results of this pilot trial, a randomized controlled trial comparing in vivo diagnosis to conventional histological assessment in matters of hospitalisation and survival will be performed.

ELIGIBILITY:
Inclusion Criteria:

Patients after haematopoietic stem cell transplantation (HSCT) who are referred to our department for clarification of one of the following symptoms:

* anorexia
* nausea
* vomiting
* abdominal pain
* diarrhoea
* intestinal bleeding

To exclude possible side effects of the conditioning therapy, GI symptoms must have occurred or persisted 20 days after the respective transplantation date [22].

Exclusion criteria:

* infection with CMV or HSV
* bacterial infection of the GI tract
* medication related symptoms
* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* refusal to participate in the study
* patient's age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
GvHD-markers on endomicroscopy | 2 years
  Establishing endomicroscopic markers of acute graft-versus-host disease in the small bowel. This outcome is a qualitative endpoint. It will be assessed descriptively.

SECONDARY OUTCOMES:
Sensitivity and Specificity of Endomicroscopy in enteral GvHD | 2 years
  At the end of the study all study derived endomicroscopic pictures will be judged by two board certified pathologists regarding presence or absence of GvHD. In comparison to the corresponding histological sections sensitivity and specificity of the technique will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Werner Dolak, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterologie and Hepatologie; Andreas Puespoek, MD, Study Director — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ferrara JL, Levine JE, Reddy P, Holler E. Graft-versus-host disease. Lancet. 2009 May 2;373(9674):1550-61. doi: 10.1016/S0140-6736(09)60237-3. Epub 2009 Mar 11. PMID 19282026
- [Background] Schulenburg A, Turetschek K, Wrba F, Vogelsang H, Greinix HT, Keil F, Mitterbauer M, Kalhs P. Early and late gastrointestinal complications after myeloablative and nonmyeloablative allogeneic stem cell transplantation. Ann Hematol. 2004 Feb;83(2):101-6. doi: 10.1007/s00277-003-0756-4. Epub 2003 Nov 13. PMID 14615909
- [Background] Nydegger A, Catto-Smith AG, Tiedemann K, Hardikar W. Diagnosis of gastrointestinal graft-versus-host disease--is rectal biopsy enough? Pediatr Blood Cancer. 2007 May;48(5):561-6. doi: 10.1002/pbc.20924. PMID 16862539
- [Background] Khan K, Schwarzenberg SJ, Sharp H, Jessurun J, Gulbahce HE, Defor T, Nagarajan R. Diagnostic endoscopy in children after hematopoietic stem cell transplantation. Gastrointest Endosc. 2006 Sep;64(3):379-85; quiz 389-92. doi: 10.1016/j.gie.2005.08.040. PMID 16923486
- [Background] Ross WA, Ghosh S, Dekovich AA, Liu S, Ayers GD, Cleary KR, Lee JH, Couriel D. Endoscopic biopsy diagnosis of acute gastrointestinal graft-versus-host disease: rectosigmoid biopsies are more sensitive than upper gastrointestinal biopsies. Am J Gastroenterol. 2008 Apr;103(4):982-9. doi: 10.1111/j.1572-0241.2007.01639.x. Epub 2007 Nov 19. PMID 18028511
- [Background] Weisdorf DJ, Snover DC, Haake R, Miller WJ, McGlave PB, Blazar B, Ramsay NK, Kersey JH, Filipovich A. Acute upper gastrointestinal graft-versus-host disease: clinical significance and response to immunosuppressive therapy. Blood. 1990 Aug 1;76(3):624-9. PMID 2378989
- [Background] Roy J, Snover D, Weisdorf S, Mulvahill A, Filipovich A, Weisdorf D. Simultaneous upper and lower endoscopic biopsy in the diagnosis of intestinal graft-versus-host disease. Transplantation. 1991 Mar;51(3):642-6. doi: 10.1097/00007890-199103000-00019. PMID 2006521
- [Background] Cruz-Correa M, Poonawala A, Abraham SC, Wu TT, Zahurak M, Vogelsang G, Kalloo AN, Lee LA. Endoscopic findings predict the histologic diagnosis in gastrointestinal graft-versus-host disease. Endoscopy. 2002 Oct;34(10):808-13. doi: 10.1055/s-2002-34257. PMID 12244503
- [Background] Thompson B, Salzman D, Steinhauer J, Lazenby AJ, Wilcox CM. Prospective endoscopic evaluation for gastrointestinal graft-versus-host disease: determination of the best diagnostic approach. Bone Marrow Transplant. 2006 Sep;38(5):371-6. doi: 10.1038/sj.bmt.1705453. PMID 16915225
- [Background] Xu CF, Zhu LX, Xu XM, Chen WC, Wu DP. Endoscopic diagnosis of gastrointestinal graft-versus-host disease. World J Gastroenterol. 2008 Apr 14;14(14):2262-7. doi: 10.3748/wjg.14.2262. PMID 18407606
- [Background] Worawattanakul S, Semelka RC, Kelekis NL, Sallah AS. MR findings of intestinal graft-versus-host disease. Magn Reson Imaging. 1996;14(10):1221-3. doi: 10.1016/s0730-725x(96)00245-7. PMID 9065914
- [Background] Kalantari BN, Mortele KJ, Cantisani V, Ondategui S, Glickman JN, Gogate A, Ros PR, Silverman SG. CT features with pathologic correlation of acute gastrointestinal graft-versus-host disease after bone marrow transplantation in adults. AJR Am J Roentgenol. 2003 Dec;181(6):1621-5. doi: 10.2214/ajr.181.6.1811621. PMID 14627585
- [Background] Klein SA, Martin H, Schreiber-Dietrich D, Hermann S, Caspary WF, Hoelzer D, Dietrich CF. A new approach to evaluating intestinal acute graft-versus-host disease by transabdominal sonography and colour Doppler imaging. Br J Haematol. 2001 Dec;115(4):929-34. doi: 10.1046/j.1365-2141.2001.03221.x. PMID 11843829
- [Background] Gorg C, Wollenberg B, Beyer J, Stolte MS, Neubauer A. High-resolution ultrasonography in gastrointestinal graft-versus-host disease. Ann Hematol. 2005 Jan;84(1):33-9. doi: 10.1007/s00277-004-0893-4. Epub 2004 Sep 1. PMID 15526100
- [Background] Yakoub-Agha I, Maunoury V, Wacrenier A, Couignoux S, Depil S, Desreumaux P, Bauters F, Colombel JF, Jouet JP. Impact of Small Bowel Exploration Using Video-Capsule Endoscopy in the Management of Acute Gastrointestinal Graft-versus-Host Disease. Transplantation. 2004 Dec 15;78(11):1697-701. doi: 10.1097/01.tp.0000141092.08008.96. PMID 15591963
- [Background] Neumann S, Schoppmeyer K, Lange T, Wiedmann M, Golsong J, Tannapfel A, Mossner J, Niederwieser D, Caca K. Wireless capsule endoscopy for diagnosis of acute intestinal graft-versus-host disease. Gastrointest Endosc. 2007 Mar;65(3):403-9. doi: 10.1016/j.gie.2005.10.042. PMID 17321239
- [Background] Schulenburg A, Kalhs P, Rabitsch W. Recommendations for diagnosis of acute gastrointestinal graft-versus-host disease in the small intestine. Transplantation. 2005 Jun 27;79(12):1767. doi: 10.1097/01.tp.0000158717.07545.ef. No abstract available. PMID 15973186
- [Background] Terdiman JP, Linker CA, Ries CA, Damon LE, Rugo HS, Ostroff JW. The role of endoscopic evaluation in patients with suspected intestinal graft-versus-host disease after allogeneic bone-marrow transplantation. Endoscopy. 1996 Oct;28(8):680-5. doi: 10.1055/s-2007-1005576. PMID 8934085
- [Background] Dolak W, Rabitsch W, Kalhs P, Wrba F, Gangl A, Haefner M. The Role of Enteroscopy in the Diagnostic Management of Acute Gastrointestinal Graft-Versus-Host Disease: A Single Centre Experience. Gastrointest Endosc 2009 Apr;69(5):AB195-6.
- [Background] Kiesslich R, Galle P, Neurath M. Atlas of endomicroscopy. Springer Medical Publishing. 2008
- [Background] Bojarski C, Gunther U, Rieger K, Heller F, Loddenkemper C, Grunbaum M, Uharek L, Zeitz M, Hoffmann JC. In vivo diagnosis of acute intestinal graft-versus-host disease by confocal endomicroscopy. Endoscopy. 2009 May;41(5):433-8. doi: 10.1055/s-0029-1214604. Epub 2009 May 5. PMID 19418398
- [Background] Epstein RJ, McDonald GB, Sale GE, Shulman HM, Thomas ED. The diagnostic accuracy of the rectal biopsy in acute graft-versus-host disease: a prospective study of thirteen patients. Gastroenterology. 1980 Apr;78(4):764-71. PMID 6986319
- [Background] Gallucci BB, Sale GE, McDonald GB, Epstein R, Shulman HM, Thomas ED. The fine structure of human rectal epithelium in acute graft-versus-host disease. Am J Surg Pathol. 1982 Jun;6(4):293-305. doi: 10.1097/00000478-198206000-00002. PMID 7051875
- [Background] Davies GR, Benson MJ, Gertner DJ, Van Someren RM, Rampton DS, Swain CP. Diagnostic and therapeutic push type enteroscopy in clinical use. Gut. 1995 Sep;37(3):346-52. doi: 10.1136/gut.37.3.346. PMID 7590429
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Dunbar KB, Okolo P 3rd, Montgomery E, Canto MI. Confocal laser endomicroscopy in Barrett's esophagus and endoscopically inapparent Barrett's neoplasia: a prospective, randomized, double-blind, controlled, crossover trial. Gastrointest Endosc. 2009 Oct;70(4):645-54. doi: 10.1016/j.gie.2009.02.009. Epub 2009 Jun 25. PMID 19559419